CLINICAL TRIAL: NCT01434303
Title: Phase I and Phase I Trastuzumab Cohort Study of Entinostat, Lapatinib and Trastuzumab in Patients With HER2-Positive Metastatic Breast Cancer in Whom Trastuzumab Has Failed
Brief Title: Entinostat, Lapatinib Ditosylate and Trastuzumab in Treating Patients With Locally Recurrent or Distant Relapsed Metastatic Breast Cancer Previously Treated With Trastuzumab Only
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03222; NCI-2011-03222 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI 8871; 2010-0842; CDR0000710891; 2010-0842 (Other: M D Anderson Cancer Center); 8871 (Other: CTEP); P30CA016672 (NIH); U01CA062461 (NIH); UM1CA186688 (NIH)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: HER2/Neu Positive; Invasive Breast Carcinoma; Recurrent Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — entinostat; Lapatinib; Trastuzumab; PF-05280014; Ogivri; trastuzumab biosimilar HLX02

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (entinostat, lapatinib ditosylate and trastuzumab) (Experimental): Patients receive entinostat PO on days 1 and 15 and lapatinib tosylate PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients in the Phase I Trastuzumab Cohort also receive maintenance dose of trastuzumab IV over 30-90 minutes every 3 weeks.
  Interventions: Drug: Entinostat; Other: Laboratory Biomarker Analysis; Drug: Lapatinib Ditosylate; Biological: Trastuzumab

INTERVENTIONS:
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lapatinib Ditosylate — Given PO
  Other Names: Tykerb
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; PF-05280014; rhuMAb HER2; RO0452317; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab-dkst

SUMMARY:
This phase I trial studies the side effects and best dose of entinostat when given together with lapatinib ditosylate and trastuzumab in treating patients with breast cancer that has spread from the original (primary) tumor to distant organs or distant lymph nodes or has recurred (come back) at or near the same place as the original (primary) tumor, usually after a period of time during which the cancer could not be detected. Entinostat and lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as trastuzumab, may interfere with the ability of tumor cells to grow and spread. Giving entinostat together with lapatinib ditosylate and trastuzumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase II dose (RP2D) for entinostat in combination with lapatinib (lapatinib ditosylate) in patients whom trastuzumab has failed for human epidermal growth factor receptor 2+ (HER2+) metastatic breast cancer (Phase I).

II. To determine the maximum tolerated dose (MTD) for entinostat in combination with lapatinib and trastuzumab in patients whom trastuzumab has failed for HER2+ metastatic breast cancer (Phase I Trastuzumab Cohort).

SECONDARY OBJECTIVES:

I. To determine the toxicity of combination therapy with entinostat and lapatinib in patients whom trastuzumab has failed for HER2+ metastatic breast cancer (Phase I).

II. To determine the toxicity of entinostat in combination with lapatinib and trastuzumab in patients whom trastuzumab has failed for HER2+ metastatic breast cancer (Phase I Trastuzumab Cohort).

EXPLORATORY OBJECTIVES:

I. Determine whether the 2-drug combination modulates the expression of HER2, phosphorylated HER2 (pHER), epidermal growth factor receptor (EGFR), phosphorylated EGFR (pEGFR), v-akt murine thymoma viral oncogene homolog 1 (Akt), and phosphorylated Akt (pAkt) in breast tumors and/or circulating tumor cells (CTCs).

OUTLINE: This is a dose-escalation study of entinostat.

Patients receive entinostat orally (PO) on days 1 and 15 and lapatinib tosylate PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients in the Phase I trastuzumab cohort also receive maintenance dose of trastuzumab intravenously (IV) over 30-90 minutes every 3 weeks.

After completion of study treatment, patients are followed up for 28 days or until toxicities are resolved.

ELIGIBILITY:
Inclusion Criteria:

* Patients have histological confirmation of invasive breast carcinoma
* Patients have locally recurrent or distant relapsed metastatic disease
* Patients have positive HER2 expression by immunohistochemistry (IHC) (3+) or fluorescence in situ hybridization (FISH) testing (> 2.0 ratio)
* Patients are able to swallow and retain oral medication (i.e., no uncontrolled vomiting, inability to swallow, or diagnosis of chronic malabsorption)
* Patients have Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must have received prior trastuzumab for > 2 month period before disease recurrence or recurrence or progression while on trastuzumab-based therapy
* Patients have ability and willingness to sign written informed consent
* Female patients of childbearing potential (a female not free from menses > 2 years or not surgically sterilized) must be willing to use an adequate barrier method of contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study; male patients who are able to father children must use an adequate barrier method of contraception
* Female patients of childbearing potential must have negative serum pregnancy test within 14 days of starting protocol therapy
* Patients with brain metastasis have no signs of progressive disease 4 months after the completion of brain metastasis treatment (radiation therapy, surgery, etc.) do not require anticonvulsants or corticosteroids, and have been off such drugs for at least 7 days
* Both men and women and members of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Patients are receiving concurrent anti-cancer therapy (chemotherapy, immunotherapy, biological therapy and hormonal therapy) while taking study medication
* Serum bilirubin >= 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >= 3 x ULN (with or without liver metastasis [mets])
* Absolute neutrophil count (ANC) < 1.5
* Hemoglobin =< 9
* Platelet =< 140,000
* Patients have an active infection and require intravenous (IV) or oral antibiotics
* Cardiac arrhythmia requiring maintenance medication
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
* Patients have a concurrent disease or condition that would make them inappropriate for study participation, or any serious medical disorder that would interfere with patients' safety
* Serum creatinine > 2.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2016-02-16 (Actual)

PRIMARY OUTCOMES:
RP2D for entinostat in combination with lapatinib ditosylate defined as the highest dose level in which 6 patients have been treated with at most 1 patient experiencing dose limiting toxicity | Up to 28 days

SECONDARY OUTCOMES:
Incidence of grade III or IV toxicities, graded according to Common Terminology Criteria for Adverse Events version 4 | Up to 28 days

OTHER OUTCOMES:
Changes in CTCs levels before and after the combination treatment of entinostat, lapatinib ditosylate and trastuzumab | Baseline up to 28 days after completion of study treatment
  Summary statistics (mean, standard deviation, median, quartiles) will be summarized for these changes in CTCs and biomarkers by patient tumor response status (yes vs. no). Changes will be compared between the two groups of patients (yes vs. no tumor response) using the two-sample t-test. If the data is skewed, Wilcoxon rank-sum test will be used.
Changes in phosphorylated Akt levels before and after the combination treatment of entinostat, lapatinib ditosylate and trastuzumab. | Baseline up to 28 days after completion of study treatment
  Summary statistics (mean, standard deviation, median, quartiles) will be summarized for these changes in CTCs and biomarkers by patient tumor response status (yes vs. no). Changes will be compared between the two groups of patients (yes vs. no tumor response) using the two-sample t-test. If the data is skewed, Wilcoxon rank-sum test will be used.
Changes in phosphorylated HER2 levels before and after the combination treatment of entinostat, lapatinib ditosylate and trastuzumab | Baseline up to 28 days after completion of study treatment
  Summary statistics (mean, standard deviation, median, quartiles) will be summarized for these changes biomarkers by patient tumor response status (yes vs. no). Changes will be compared between the two groups of patients (yes vs. no tumor response) using the two-sample t-test. If the data is skewed, Wilcoxon rank-sum test will be used.
Changes in phosphorylated EGFR levels before and after the combination treatment of entinostat, lapatinib ditosylate and trastuzumab | Baseline up to 28 days after completion of study treatment
  Summary statistics (mean, standard deviation, median, quartiles) will be summarized for these changes biomarkers by patient tumor response status (yes vs. no). Changes will be compared between the two groups of patients (yes vs. no tumor response) using the two-sample t-test. If the data is skewed, Wilcoxon rank-sum test will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Naoto T Ueno, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States